CLINICAL TRIAL: NCT03207087
Title: WEB® Intrasaccular Therapy Study China Clinical Trial Protocol
Brief Title: The WEB®-IT China Clinical Study
Acronym: WEB-IT China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-16-001
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Wide Neck Bifurcation Intracranial Aneurysms

STUDY DESIGN:
Intervention Model Description: Single group assignment
Masking Description: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- WEB Aneurysm Embolization Device (Experimental): The WEB is an intra-aneurysmal device intended for use in endovascular embolization of intracranial aneurysms. The intended therapeutic effect of the WEB device is to line the neck of the aneurysm with a metallic structure that disrupts the inflow of blood, causing hemostasis within the aneurysm sac, and leading to thrombus formation within the implant. Subjects will be screened for study eligibility after giving informed consent.
  Interventions: Device: WEB Aneurysm Embolization

INTERVENTIONS:
Device: WEB Aneurysm Embolization — Subjects will be screened for study eligibility after giving informed consent. The WEB embolization procedure will be performed in the catheterization room using standard angiographic techniques.

SUMMARY:
This trial is a prospective, multicenter, single-arm confirmatory clinical trial. The study is to confirm the safety and effectiveness of the WEB Aneurysm Embolization System demonstrated in the US WEB-IT Study for the treatment of intracranial wide-neck bifurcation aneurysms. The study's primary endpoints include a primary effectiveness endpoint and a primary safety endpoint. The study device must meet both endpoints. The primary effectiveness endpoint is adjudicated by an independent third party core lab.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 and ≤75 years old
* Patient must have a single ruptured or unruptured IA(intracranial aneurysm)requiring treatment
* Patient must sign and date IRB/EC approved written informed consent prior to initiate of any study procedures

Exclusion Criteria:

* Patient has an IA with characteristics unsuitable for endovascular treatment
* Patient has stroke-in-evolution within the prior 60-days
* Patient has had an SAH(subarachnoid hemorrhage) from a nonindex IA or any other intracranial hemorrhage within 90 days
* Patient's index IA was previously treated
* Patient is pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint: Complete (angiographic) aneurysm occlusion as assessed by Core Lab, without parent artery stenosis | 12 month
  Proportion of complete (angiographic) aneurysm occlusion as assessed by Core Lab without retreatment, recurrent subarachnoid hemorrhage, without significant parent artery stenosis (>50% stenosis) at one year after treatment.
Primary Safety Endpoint: Proportion of death and major stroke | 12 month
  Proportion of death of any nonaccidental cause or any major stroke (defined as an ischemic or hemorrhagic stroke resulting in an increase of 4 points or more on the National Institutes of Health Stroke Scale) within the first 30 days after treatment or major ipsilateral stroke or death due to neurologic cause from day 31 to the 1 year after treatment.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Changhai Hospital Affiliated to The Second Military Medical University ( Shanghai Changhai Hospital), Shanghai, Shanghai Municipality
  - West China, Chengdu, Sichuan
  - Tiantan Hospital, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - The Second affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Huashan Hospital, Shanghai
  - The General Hospital of Shenyang Military, Shenyang
  - Tangdu Hospital, the Fourth Military Medical University, Xi'an

REFERENCES:
- [Derived] He C, Xu J, Gao X, Li G, Liang G, Jun Y, Zhao Z, Fang B, Xie X, Liu A, Zhang J, Zhang H, Liu J. Woven EndoBridge intrasaccular therapy for the treatment of unruptured wide-necked bifurcation aneurysms: a prospective study in a Chinese population. Chin Neurosurg J. 2026 Jan 20;12(1):2. doi: 10.1186/s41016-025-00418-2. PMID 41559830